CLINICAL TRIAL: NCT07063056
Title: Curcumin and Astaxanthin for Lowering Triglyceride Readings and Inflammation
Brief Title: Curcumin & Astaxanthin for Lowering Triglyceride Readings and Inflammation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medinutra LLC (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: TgStudy
Record Dates: First submitted 2025-07-03; First posted 2025-07-14 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2025-07

CONDITIONS: Triglycerides
Keywords: Triglycerides; Antioxidants; Inflammation
MeSH Terms: conditions — Inflammation | interventions — Curcumin; astaxanthine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Control (Placebo Comparator): Subjects will be given 1 capsule per day of a small amount of cellulose
  Interventions: Other: Placebo Control
- Regular dose curcumin (Experimental): Subjects will be given 1 capsule per day of a typical amount of Longvida curcumin (80 mg curcumin)
  Interventions: Dietary Supplement: Curcumin (Longvida™)
- Low dose curcumin (Experimental): Subjects will be given 1 capsule per day of 40 mg curcumin which is half the typical amount of Longvida curcumin
  Interventions: Dietary Supplement: Half Dose Curcumin (Longvida™)
- Astaxanthin (Experimental): Subjects will be given 1 capsule per day of a typical amount of astaxanthin (12 mg curcumin)
  Interventions: Dietary Supplement: Astaxanthin

INTERVENTIONS:
Dietary Supplement: Curcumin (Longvida™) — 1 capsule per day at a usual curcumin dose for this particular product (80 mg curcumin)
  Arms: Regular dose curcumin
Dietary Supplement: Half Dose Curcumin (Longvida™) — 1 capsule per day at half the usual curcumin dose for this particular product (40 mg curcumin as the half dose)
  Arms: Low dose curcumin
Dietary Supplement: Astaxanthin — 1 capsule per day at a usual astaxanthin dose (12 mg)
  Arms: Astaxanthin
Other: Placebo Control — Subject will get 1 capsule per day of a small amount of cellulose
  Arms: Control

SUMMARY:
Two dietary supplements are each being compared to a placebo for the ability to help maintain triglycerides in the normal range. The subjects will be adult men and women with moderately high TG values. Serum triglycerides will be measured before and after 6 weeks of taking 1 capsule per day of either Longvida Curcumin, astaxanthin, or a placebo. A few side blood analysis will also be done. These measures are relevant to low level inflammation.

DETAILED DESCRIPTION:
Background Moderately high readings for serum TG have been thought to place many people at risk for cardiovascular disease (CVD) and other problems. However, for a few years, doubts were expressed about high TG as an independent risk factor for CVD and maybe other problems in most people. More recently, the tide has begun to turn back due to new studies and new attention to old studies. Now, TG readings are again being thought to affect vulnerability to CVD, fatty liver, high blood sugar, and other problems including general inflammation. Some of these studies have shown evidence that TG effects can be independent of LDL or total cholesterol readings. Also, one of these studies suggest that even dropping TG readings from the top of the normal range to lower values can produce benefits.

People with TG readings between the top of the normal range to moderately high usually do not take drugs to lower TG values. Therefore, a need exists for cost effective, low side effect alternatives to help maintain normal TG readings. Nutritional supplements could fit in here. The Dietary Supplement and Education Act (DSHEA) allows for structure function claims of helping maintain blood lipids in the normal range. Low level general inflammation, which falls below what's seen with inflammatory diseases or injury, can also raise the risk for many health problems. Drugs are not generally employed to minimize this type of inflammation. So, as with moderately high TG readings, relatively safe and inexpensive non-drug alternatives can be sought (including nutritional supplements).

This researcher has found that under certain conditions, two natural ingredients each lower TG readings. One ingredient is a high absorption form of curcumin extract from the spice turmeric (Longvida Optimized Curcumin®). A dose of 400 mg per day (80 mg curcumin) lowered TG levels in healthy middle aged women. Aanother group has found that a third ingredient, astaxanthin can produce a substantial drop in TG values. A dose of 12 mg/day was more effective than 6 mg but the same as 18 mg. Also of note, readings for HDL cholesterol, the so called good cholesterol, rose a little. Another astaxanthin study found a drop in TG values in people with type 2 diabetes. A TG lowering effect of astaxanthin has also been seen in animal studies.

It's doubtful that any of these three ingredients could produce the really large TG drops needed by people with very high values. Even so, for people in the borderline to moderately high range, these ingredients, especially in combination, could help maintain normal range values.

Eventually, a combination product could be made of astaxanthin + Longvida Optimized Curcumin® + the third ingredient. However, there is work to be done before that can be considered. One lacking is that three ingredients have never been tried in combination. But, even before trying that, another issue must be addressed. For all three ingredients, the human research cited above have all been done in subjects whose TG readings were good to begin with. Therefore, it is not known how these ingredients, combined or individually, will affect TG readings in people with higher starting values.

On the inflammation side, both curcumin and astaxanthin are considered anti-inflammatory though a lot of disjointed data exists. A meta analysis exists for supplementation of curcumin and supplementation of astaxanthin in relation to c-reactive protein (CRP), a general marker of inflammation. Each analysis concluded that overall, CRP was decreased. However, some inconsistency existed in terms of results, types of subjects examined, doses, exact nature of the extracts, and co-treatments. The latter hold particular importance for curcumin, which was sometimes given with piperine, which can conceivably have its own effects (good and bad). Thus, a need exists to study this project's type of curcumin and astaxanthin at reasonable doses in a fairly broad population.

One possible anti-inflammatory mechanism of both astaxanthin and curcumin is elevation of body glutathione. This molecule can inhibit inflammation. This project will examine whole blood glutathione.

One body area where inflammation protection may be especially useful is the liver. Both curcumin and astaxanthin have shown protection against chemically induced liver injury in experimental animals. In addition, turmeric, the source of curcumin, has been used in Indian traditional medicine for treating liver problems. This researcher has found that in generic middle aged women without liver problems, Longvida lowered readings for alanine amino transferase or ALT. ALT is not a direct indicator of inflammation. However, liver inflammation can cause liver cell damage which leaks ALT into serum to elevate readings. The results obtained by this investigator need to be extended.

Hypothesis This proposed project tests the hypothesis that astaxanthin or Longvida supplementation will lower TG readings in people with normal to moderately high starting values. A secondary hypothesis is that the supplementation will raise HDL cholesterol readings and depress values for some markers of low level inflammation.

Methods Subjects will be adult males and females aged 21-59 that lack unstable health problems that can affect TG or systemic inflammation readings. Subjects in this project will have starting TG reading of 140-250 mg/dL. Initially, this eligibility will be based on eligibility questionnaire. However, if the initial blood draw finds TG readings outside the range, subjects will be excluded and replaced. Other discontinuations will be for a subject's decision or a change in health or medication disclosed by the subject to Medinutra. For these discontinuations, subjects will not be replaced. In the applicant's experience, no dropouts, or at most one, would be expected for this type of study.

For 6 weeks, subjects will take one of the following orally as one capsule/day (up to16 people/group):

Placebo (cellulose at a low dose) Astaxanthin at 12 mg/day-from BGG Longvida Optimized Curcumin® at 400 mg per day (80 mg curcumin)-from Verdure Sciences Longvida Optimized Curcumin® at 200 mg per day (40 mg curcumin)-from Verdure Sciences

The 80 mg curcumin dose is a standard amount for this product. The 40 mg dose is being tried as a step to determining the lowest dose that can produce benefits. The astaxanthin amount is based on a dose response study for TG effects. Blood will be drawn before and after the intervention by a Labcorp facility near the subjects' residence. Labcorp will do all the study analysis on the blood samples.

Neither Labcorp nor the study subjects will not know the assigned capsule identity. Thus, this will be double blinded and randomized in terms of the participants and analyzers

For each measure, for each of the treatment groups, pre- and post-treatment values will be compared by paired t-test. In addition, the changes in values for each supplement group will be compared to placebo by unpaired t-test. For non-normal distribution, nonparametric tests can be used. Also, each group will be compared to the others by ANOVA followed by Tukey analysis when applicable. Significance is set at p < 0.05 for all tests.

Subject numbers and power calculation This project is intended to see if further research is justified on certain wellness parameters in response to each of two supplements. Further research would be on the individual ingredients as well as the combination of both ingredients as well as these two ingredient + another ingredient. Justification for more work will only occur if substantial changes occur consistently. Therefore, a relatively small subject number should be sufficient to see such patterns. A power calculation was done for changes in serum TG levels for Longvida vs placebo. A previous study from this researcher got a 15% drop in people with low starting values. The percent change may be bigger in people with higher starting values, but the power calculation was done with 15%. Placebo was set at 2%. An upper end of SD for the changes is hypothesized at 8.5%. Using a power value of 0.95 and p = 0.01, 15 subjects are needed per group. Recruitment will shoot for 16 subjects to allow for 1 drop out per group. Dropouts should not occur much if at all. That's because participation is not demanding and subjects can't tell if a treatment is not "working."

Safety considerations. A safety review of astaxanthin says that natural versions are safe at doses equal or greater than the current project dose. This was based on 35 human studies. The FDA classifies curcumin as Generally Regarded as Safe (GRAS). The dose there is less than the higher dose in the current project, but only by 25%.

Despite this classification, and despite use of curcumin to treat liver problems, a few reports of curcumin-induced liver injury have been reported. To my knowledge, none have involved the form or dose of the current project. A survey was done on liver toxicity cases where a person was taking supplements of either curcumin or turmeric, the spice that contains curcumin. In 12 years, only 10 cases were found. The authors of the survey concede that not all the cases of liver toxicity could be definitely attributed to curcumin or turmeric.

ELIGIBILITY:
Inclusion Criteria:

* Triglyceride reading of 140-250 mg/dL
* Age 21-59

Exclusion Criteria:

* Uncontrolled diabetes
* Hypothyroidism or other hormonal problems that have not stabilized
* Any liver diseases being actively treated
* Cancer
* Renal dialysis use
* Rheumatoid arthritis and related issues like lupus
* Inflammatory bowel disease
* Smoking
* Low blood pressure
* Having more than 5 alcoholic drinks per week
* Extreme obesity (BMI over 37)
* Pregnancy or lactation

Ages: 21 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 64 (Estimated)
Dates: Start 2025-07-18 (Actual); Primary Completion 2025-11-15 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Trilgycerides | Pre and post 6 week intervention
  Serum triglyceride readings (mg/dL)

SECONDARY OUTCOMES:
Other blood lipids | Before and after the 6 week intervention
  Serum values for commonly measured blood measures for comparison purposes: total cholesterol (mg/dL, LDL cholesterol (mg/dL), and HDL cholesterol (mg/dL) These are not expected to be affected by the interventions except possibly a small rise in HDL cholesterol post-intervention in some groups.
Inflammation markers | Measures will be from blood samples taken before and after the 6 week intervention.
  As a secondary consideration, this study will assess 3 blood measures relevant to low level inflammation: serum c reactive protein (mg/dL), serum alanine aminotransferase (ALT-Units/L), and whole blood glutathione (mg/L)

CONTACTS AND LOCATIONS:
Overall Officials: Robert DiSilvestro, Ph.D., Principal Investigator — Medinutra LLC
Locations (1):
- Medinutra LLC, Dublin, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] DiSilvestro RA, Joseph E, Zhao S, Bomser J. Diverse effects of a low dose supplement of lipidated curcumin in healthy middle aged people. Nutr J. 2012 Sep 26;11:79. doi: 10.1186/1475-2891-11-79. PMID 23013352
- [Background] Tikhonoff V, Casiglia E, Virdis A, Grassi G, Angeli F, Arca M, Barbagallo CM, Bombelli M, Cappelli F, Cianci R, Cicero AFG, Cirillo M, Cirillo P, Dell'oro R, D'elia L, Desideri G, Ferri C, Galletti F, Gesualdo L, Giannattasio C, Iaccarino G, Mallamaci F, Maloberti A, Masi S, Masulli M, Mazza A, Mengozzi A, Muiesan ML, Nazzaro P, Palatini P, Parati G, Pontremoli R, Quarti-Trevano F, Rattazzi M, Reboldi G, Rivasi G, Russo E, Salvetti M, Temporelli PL, Tocci G, Ungar A, Verdecchia P, Viazzi F, Volpe M, Borghi C. Prognostic Value and Relative Cutoffs of Triglycerides Predicting Cardiovascular Outcome in a Large Regional-Based Italian Database. J Am Heart Assoc. 2024 Feb 6;13(3):e030319. doi: 10.1161/JAHA.123.030319. Epub 2024 Jan 31. PMID 38293920
- [Background] Kraaijenhof JM, Stroes ESG. Inflammatory Effects of Triglycerides: Relevant or Redundant? JACC Basic Transl Sci. 2023 May 22;8(5):476-478. doi: 10.1016/j.jacbts.2023.04.005. eCollection 2023 May. PMID 37325399
- [Background] Yoshida H, Yanai H, Ito K, Tomono Y, Koikeda T, Tsukahara H, Tada N. Administration of natural astaxanthin increases serum HDL-cholesterol and adiponectin in subjects with mild hyperlipidemia. Atherosclerosis. 2010 Apr;209(2):520-3. doi: 10.1016/j.atherosclerosis.2009.10.012. Epub 2009 Oct 14. PMID 19892350

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-05-16): https://cdn.clinicaltrials.gov/large-docs/56/NCT07063056/Prot_SAP_000.pdf